CLINICAL TRIAL: NCT01000038
Title: Wii-fit for Activity, Balance and Gait in Assisted Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0085-09-FB
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Falls; Alzheimer's Disease
Keywords: Wii-Fit; Assisted living; Alzheimer's dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wii-Fit Intervention (Experimental): Intervention: Subjects in this arm participate in Wii-Fit exercises
  Interventions: Other: Wii-Fit intervention; Other: Walking
- Walking Intervention (Active Comparator): Intervention: Subjects in this arm participate in walking
  Interventions: Other: Walking

INTERVENTIONS:
Other: Wii-Fit intervention — Half hour daily, 5 days a week for 8 weeks
  Other Names: Exercise intervention
  Arms: Wii-Fit Intervention
Other: Walking — Half hour daily, five days a week for 8 weeks
  Other Names: Exercise intervention

SUMMARY:
Falls in Alzheimer's Disease (AD) are common and lead to fractures, acute hospitalizations and increased rate of institutionalization. Poor balance and gait abnormalities, commonly associated with AD, are risk factors. Improving balance and gait abnormalities is critical in preventing these falls. Walking is the most commonly recommended home-based exercise program for elderly by primary care providers. However, it is difficult to engage patients with AD in long term exercise programs. Barriers include lack of motivation, poor engagement, and external factors such as the cost of physical therapy (PT).

The use of readily available technology might bridge this gap by providing high level of engagement via use of multimedia at an affordable price. Wii-Fit is a Nintendo gaming console used for aerobics, strength training, and balance activities. It is a TV based self-directed activity where virtual trainers talk the user through the activity while tracking progress. Some skilled nursing facilities have started using the Wii-Fit as an adjunct to PT and note improvement in balance along with social benefits, but no systematic studies are done to generalize the findings. This study will compare changes in balance and daily living activities between a group receiving Wii-Fit training and another receiving a walking exercise program.

DETAILED DESCRIPTION:
Purpose of the study: Falls in Alzheimer's Disease (AD) are common and lead to fractures, acute hospitalizations and increased rate of institutionalization. Poor balance and gait abnormalities, commonly associated with AD, are risk factors for falls. Improving balance and gait abnormalities is critical to prevent falls in AD.

Exercise interventions improve gait and balance in elderly. Walking is the most commonly recommended home-based exercise program for elderly by primary care providers. However, it is difficult to engage patients with AD in long term exercise programs. Barriers to exercise programs include lack of motivation, poor engagement, and external factors such as the cost of physical therapy (PT). Use of readily available technology might bridge this gap by providing high level of engagement via use of multimedia at an affordable price.

Wii-Fit is a Nintendo gaming console used for aerobics, strength training, and balance activities. This device includes a balance board that senses weight, movement and balance. Wii-Fit is a TV based self-directed activity not limited by the constraint of a therapist's presence. Virtual trainers talk the user through the activity while tracking progress. Furthermore, visual and auditory feedback improves engagement. Some skilled nursing facilities have started using the Wii-Fit as an adjunct to PT, and note improvement in balance along with social benefits but no systematic studies are done to generalize the findings.

The investigators propose an 8 week prospective randomized study with the treatment group receiving the exercise program delivered by Wii-Fit system and the comparison arm receiving a walking exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60
* Alzheimer's Dementia, mild (MMSE ≥ 18)
* Residing in assisted living facility
* Presence of legal surrogate

Exclusion Criteria:

* History of myocardial infarction, TIA or stroke in last 6 months
* Presence of serious mental illness impacting memory
* Active cancer except skin cancer
* Medical conditions likely to compromise survival (e.g. severe congestive heart failure)
* Severe sensory and musculoskeletal impairments
* Using wheel-chair

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03-30 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 8 weeks
  Balance test

SECONDARY OUTCOMES:
Activities of Daily Living | 8 weeks
  Daily functioning test
Instrumental Activities of Daily Living | 8 weeks
  Higher level of functioning assessment
Timed Up and Go | 8 weeks
  Functional performance test
Quality of Life-AD | 8 weeks
  Global quality of life measure
Mini Mental State Exam | 8 weeks
  Global cognitive screen
Actigraphy | 3 days before the intervention and 3 days during the intervention
  Activity measure
Trails A and B | 8 weeks
  Executive function measure

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana P Padala, MD, MS, Principal Investigator — University of Nebraska
Locations (1):
- Parson's House Assisted Living, Omaha, Nebraska, United States

REFERENCES:
- [Result] Padala KP, Padala PR, Malloy TR, Geske JA, Dubbert PM, Dennis RA, Garner KK, Bopp MM, Burke WJ, Sullivan DH. Wii-fit for improving gait and balance in an assisted living facility: a pilot study. J Aging Res. 2012;2012:597573. doi: 10.1155/2012/597573. Epub 2012 Jun 13. PMID 22745909